CLINICAL TRIAL: NCT07268846
Title: Randomized Clinical Trial on the Use of Preoperative Postbiotic Supplementation in Colorectal Cancer Surgery
Brief Title: Use of Preoperative Postbiotic Supplementation in Colorectal Cancer Surgery
Acronym: POSBIO-CRC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: AC Camargo Cancer Center (Other)
Responsible Party: Principal Investigator, Samuel Aguiar Jr, MD, PhD, Head of Colorectal Cancer Reference Center at A.C.Camargo Cancer Center, AC Camargo Cancer Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: CEP3592/24
Record Dates: First submitted 2025-11-17; First posted 2025-12-08 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-12

CONDITIONS: Cancer (Colon Cancer, Breast Cancer, Lymphoma, Chronic Lymphoma Leukemia, Multiple Myeloma)
Keywords: Colorectal cancer surgery; Postbiotic; colorectal cancer; intestinal microbiota; nutritional intervention; inflammation
MeSH Terms: conditions — Neoplasms; Colonic Neoplasms; Breast Neoplasms; Lymphoma; Multiple Myeloma; Colorectal Neoplasms; Inflammation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Placebo group (Placebo Comparator): Participants will receive three oral capsules per day, containing no active substance and identical in appearance to the study capsules, for seven consecutive days.
  Interventions: Other: Placebo
- Oral postbiotic supplementation ( Butyrate) (Experimental): The formulation will contain tributyrin as the active compound, which acts directly on the large intestine. Tributyrin serves as a source of butyrate, a short-chain fatty acid. Total daily dose of 900 mg, divided into three 300 mg capsules, for seven consecutive days.
  Interventions: Dietary Supplement: Postbiotic

INTERVENTIONS:
Dietary Supplement: Postbiotic — Butyrate directly influences the gastrointestinal microbiota and exhibits potent anti-inflammatory effects by locally inhibiting inflammatory mediators in the intestinal epithelium, thereby enhancing mucosal barrier integrity. It also mitigates excessive inflammation through the modulation of immune cells, promoting the activity of M2 macrophages and regulatory T cells.
  Furthermore, butyrate is thought to modulate intestinal receptor hypersensitivity, leading to reduced intraluminal pressure and improved peristaltic function. This mechanism may underlie its therapeutic role in clinical conditions associated with diarrhea and in preventing the loss of water, sodium, chloride, and potassium.
  Arms: Oral postbiotic supplementation ( Butyrate)
Other: Placebo — Participants will receive three oral capsules per day, containing no active substance and identical in appearance to the study capsules, for seven consecutive days.
  Arms: Placebo group

SUMMARY:
The treatment of colorectal cancer, in the absence of metastases, is primarily based on surgical removal. Colorectal surgery, which involves resecting part of the intestine and restoring intestinal continuity, carries a risk of complications. This study aims to evaluate whether oral supplementation with a postbiotic at a dose of 900 mg for 7 days prior to surgery reduces the rate of postoperative complications.

DETAILED DESCRIPTION:
Recent studies have underscored the influence of gut microbiota composition on the incidence of postoperative complications following intestinal surgery. Microorganisms naturally present in the intestinal environment produce a variety of substances that may exert either beneficial or detrimental effects on human health. Emerging evidence indicates a protective role for metabolites derived from these microorganisms.

Pharmacological modulation of these metabolites for human supplementation has led to the development of postbiotics. Recent research has demonstrated that certain postbiotics, particularly short-chain fatty acids such as butyrate, possess immunomodulatory properties and contribute to maintaining the integrity of the intestinal barrier in inflammatory bowel disease.

This study will include two groups of participants: one group will receive a daily supplementation of 900 mg of butyrate, while the other will receive a placebo, for seven days prior to surgery. A total of 164 participants are expected to be enrolled, and the study will be conducted over a two-year period.

The present proposal aims to assess the effectiveness of a postbiotic in reducing postoperative complications in colorectal cancer surgery, with an anticipated 50% reduction in the overall postoperative complication rate in the intervention arm. If confirmed, such a reduction would represent a substantial decrease in morbidity and healthcare costs throughout the treatment pathway for this specific population.

ELIGIBILITY:
Inclusion Criteria:

* Individuals diagnosed with malignant neoplasm of the large intestine, specifically adenocarcinoma.
* Patients over 18 years of age, of both sexes.
* Patients who agree to participate in the study and sign the informed consent form.

Exclusion Criteria:

* Emergency or urgent surgeries.
* Cytoreductive surgeries involving intraoperative intraperitoneal chemotherapy.
* Extended surgeries for the treatment of recurrent tumors.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 164 (Estimated)
Dates: Start 2025-06-01 (Actual); Primary Completion 2027-06-01 (Estimated); Study Completion 2027-06-01 (Estimated)

PRIMARY OUTCOMES:
Postoperative complications within 30 days (Clavien-Dindo grade II or higher) | 30 days after colorectal cancer surgery
  Clinical or surgical postoperative complication - Clavien-Dindo grade II or higher .

SECONDARY OUTCOMES:
C-reactive protein (CRP) levels after surgery | Baseline (within 7 days before surgery) and postoperative day 3
  Serum C-reactive protein (CRP) concentration (mg/L) measured preoperatively (within 7 days before surgery) and on postoperative day 3. The primary comparison will be the CRP level on postoperative day 3 between the postbiotic and control groups, as well as the change in CRP from baseline to postoperative day 3.
Gastrointestinal postoperative complications (Clavien-Dindo grade II or higher) | 30 days after surgery
  Gastrointestinal postoperative complication : Clavien-Dindo grade II or higher within 30 days after colorectal cancer surgery (including, for example, prolonged postoperative ileus, bowel subocclusion or obstruction, anastomotic leakage, enteric fistula, intra-abdominal abscess, or gastrointestinal bleeding requiring intervention).
Nutritional status and body composition assessed by preoperative computed tomography | Baseline (preoperative CT scan performed within 8 weeks before surgery); postoperative complications assessed within 30 days after surgery
  Preoperative body composition assessment will be performed using abdominal computed tomography scans obtained for colorectal cancer staging. Skeletal muscle area at the level of L3, skeletal muscle index (SMI), and visceral adipose tissue area will be quantified. The prevalence of sarcopenia, visceral obesity, and sarcopenic obesity will be described, and the associations between these body composition phenotypes and postoperative complications within 30 days will be explored.
Dietary intake assessment using a Food Frequency Questionnaire (FFQ) | Baseline (preoperative assessment); postoperative complications assessed within 30 days.
  Habitual dietary intake will be assessed preoperatively using a validated Food Frequency Questionnaire (FFQ). Associations between identified dietary intake patterns and postoperative complications within 30 days will be explored, as well as potential interactions between habitual diet and the response to preoperative postbiotic supplementation.

CONTACTS AND LOCATIONS:
Overall Officials: Samuel A Junior, MD, PhD, Principal Investigator — A.C.Camargo Cancer Center
Locations (1):
- A.C.Camargo Cancer Center, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No